CLINICAL TRIAL: NCT02843581
Title: Combination of Cryosurgery and NK Immunotherapy for Advanced Esophageal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fuda Cancer Hospital, Guangzhou (Other)
Collaborators: Shenzhen Hank Bioengineering Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NK-esopha
Record Dates: First submitted 2016-07-16; First posted 2016-07-26 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2019-07

CONDITIONS: Metastatic Esophageal Cancer
Keywords: Esophageal Cancer; NK immunotherapy; Safety; Efficacy
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Cryosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cryosurgery and NK immunotherapy (Experimental): We use comprehensive cryosurgery to destroy big tumors, and use multiple (more than 6 times) NK immunotherapy to destroy small tumors
  Interventions: Device: Cryosurgery; Biological: NK immunotherapy
- Cryosurgery (Active Comparator): We use comprehensive cryosurgery to destroy big tumors
  Interventions: Device: Cryosurgery

INTERVENTIONS:
Device: Cryosurgery — Argon-helium cryosurgical system
Biological: NK immunotherapy — Nutral killer cell immunotherapy for more than 6 times
  Arms: Cryosurgery and NK immunotherapy

SUMMARY:
The aim of this study is the safety and efficacy of cryosurgery plus NK immunotherapy to advanced esophageal cancer.

DETAILED DESCRIPTION:
By enrolling patients with pancreatic cancer adapted to enrolled criteria, this study will document for the first time the safety and the short and long term efficacy of the combined therapy using cryosurgery and nature killer (NK) cells for advanced esophageal cancer.

The safety will be evaluated by statistics of adverse reactions.The efficacy will be evaluated according to local relief degree, progress free survival (PFS) and overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* All standard therapies have failed according to NCCN guidelines or the patient refuses standard therapies after cancer recurrence
* Body tumor 1-6, the maximum tumor length < 5 cm
* KPS ≥ 70, lifespan > 6 months
* Platelet count ≥ 80×109/L，white blood cell count ≥ 3×109/L, neutrophil count ≥ 2×109/L, hemoglobin ≥ 80 g/L

Exclusion Criteria:

* Patients with cardiac pacemaker
* Patients with brain metastasis
* Patients with grade 3 hypertension or diabetic complication, severe cardiac and pulmonary dysfunction

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Relief degree | 3 months
  It will be evaluated by the Response Evaluation Criteria in Solid Tumors（RECIST）

SECONDARY OUTCOMES:
Progress free survival（PFS） | 1 year
Overall survival（OS） | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Guifeng Liu, PhD, Principal Investigator — Fuda Cancer Hospital, Guangzhou
Locations (1):
- Fuda cancer institute in Fuda cancer hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes